CLINICAL TRIAL: NCT04444115
Title: Loneliness During the COVID-19 Pandemic: Change and Predictors of Change From Strict to Lifted Social Distancing Protocols
Brief Title: Loneliness During Strict and Lifted Social Distancing Protocols Against the COVID-19 Pandemic
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Modum Bad (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Principal Investigator, Asle Hoffart, Prof, Modum Bad
Other Study IDs: 802810-1
Record Dates: First submitted 2020-06-20; First posted 2020-06-23 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Loneliness During COVID-19
Keywords: COVID-19, social distancing, loneliness, worry, rumination, depression, anxiety
MeSH Terms: conditions — COVID-19; Rumination Syndrome; Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Description The aim of the present study is to investigate (a) changes in the levels of loneliness in the general adult population from a period of strict distancing protocols designed to impede transmission of the corona virus (T1) to a later period of lifted distancing protocols period (T2), (b) the risk and resilience factors for persistence in loneliness across these periods and (c) the associations between loneliness at T1 and changes in loneliness from T1 to T2 and changes in psychopathology symptoms from T1 to T2.

An investigation of loneliness persistence in addition to its association with risk factors and the persistence of psychopathology provides a knowledge basis for employing interventions that protect the general public against increased distress and dysfunction during and after society's handling of pandemics.

DETAILED DESCRIPTION:
Hypotheses and research questions:

The hypotheses (Hs) and explorative research questions of the present study were:

H1: The lifting of the social distancing protocols are associated with decreased loneliness. Exploratory question 1. What is the proportion showing a reliable change in loneliness? Exploratory question 2. What are the associations of the stable (demographic) factors age, gender, educational level, civil status, employment status, psychiatric diagnosis status and refugee status with change in loneliness from T1 to T2? H2: Of psychological factors, higher level at T1 and less reduction from T1 to T2 in worry about job and/or economy, worry about health (health anxiety), maladaptive mental and behavioral coping, and negative and positive metacognitions will be associated with less reduction in loneliness from T1 to T2, above and beyond the influence of pre-existing stable risk factors.

Explorative question 3. What are the potential protective effects of doing new positive activities at home, experiencing nature and performing aerobic physical exercise? That is, is higher level at T1 and more increase from T1 and T2 of these activities related to more reduction of loneliness from T1 to T2? H3: More loneliness at T1 will be associated with less reduction of depressive and anxiety symptoms from T1 to T2. Less reduction in loneliness from T1 to T2 will be associated with less reduction of symptoms in the same time frame. Because variables related to loneliness may confound the relationship between loneliness and psychopathology symptoms, the variables showing significant associations for Hypothesis 2 and 3 will be controlled for. However, psychiatric diagnosis will not be included as a control variable because T1 level of depression and anxiety symptoms is controlled.

Study design and participants The design is a longitudinal observational survey of the general adult Norwegian population during the COVID-19 pandemic. Eligible participants are all individuals of 18 years and above, who are living in Norway and thus experience identical distancing protocols, and who provide informed consent to participate in the study. The strict distancing protocols were implemented in Norway at March 12. 2020 and the first data collection in this period has already been done. It lasted seven days and was between March 31st 2020 and April 7th 2020. Thus, the strict protocols had been held constant during the two weeks prior to data collection, as well as during the data collection week. Furthermore, no new information was given by the government during this period with regard to changes of distancing protocols, keeping expectation effects constant. From June 15., the majority of the strict distancing protocols will be lifted in Norway, and lifted distancing protocol period is defined from this date. Data are set to be collected from the sample providing data in the first collection (N = 10 084), starting one week after the lifting data, that is, from 22th of June. The collection will last until enough data has been collected, but no longer than three weeks.

Ethical approval of the study was granted by The Regional Committee for Medical and Health Research Ethics and the Norwegian Centre for Research Data (reference numbers: 125510 and 802810, respectively, where the study protocol and analysis plan was approved prior to data collection. The study is conducted in accordance with the guidelines of the Strengthening the Reporting of Observational Studies in Epidemiology statement (STROBE; Von Elm et al., 2007). The pre-registered protocol for a study of loneliness based on the first T1 data collection can be found at Clinicaltrials.gov (Identifier: NCT04365881). The study is part of The Norwegian COVID-19, Mental Health and Adherence Project (Ebrahimi, Hoffart, & Johnson, 2020).

Procedures The survey was disseminated online in a systematic manner to give the adult population an equal opportunity to participate in the study. The dissemination procedure involved information about the survey through broadcasting on national, regional, and local news channels and provision of the online survey to a random selection of Norwegian adults on Facebook. The dissemination procedure is described in detail elsewhere (Ebrahimi et al., 2020).

The stopping rule for the first data collection was designed to ensure that the social distancing protocols were held constant for two weeks prior to and the week during the data collection period, as well as controlling for expectation effects by stopping data collection instantly once information concerning forthcoming modification of the protocols were given. The second data collection will start one week after the social distancing protocols are lifted (June 22.) and last three weeks.

Inference criteria Given the large sample size in this study, the investigators pre-define their significance level: p < 0.001 to determine significance.

Sample size and power The sample size T1 included 10 084 participants, ascertaining power for the questions asked. For the present study, all these participants will be invited to participate at T2 in accordance with the study plan.

Statistical analyses Repeated surveys like the present one typically have a lot of drop out and missing data. Therefore, we will use mixed models instead of paired t-tests, repeated measures ANOVAs, and ordinary least square regression to analyze the data. Mixed models use maximum likelihood estimation, which is the state of the art approach to handle missing data (Schafer & Graham, 2002). Especially if data are missing at random, which is likely in our survey, mixed models give more unbiased results than the other analytic methods (O'Connel et al., 2017).

In preliminary analyses, and for each of the dependent variables (ULS-8, PHQ-9, GAD-7), the combination of random effects and covariance structure of residuals that gives the best fit for the "empty" model (the model without fixed predictors except the intercept) will be chosen. Akaike's Information Criterion (AIC) will used to compare the fit of different models. Models that give a reduction in AIC greater than 2 will be considered better (Burnham & Anderson, 2004). The program SPSS 25.0 will be used (IBM Corp, 2018).

First, H1 about decrease in ULS-8 will be tested by using ULS-8 as dependent variable in a model using time (T1 = 0, T2 = 1) as a predictor. Second, demographic group variables will be added as predictors. Third, the T1 levels of worry about job and/or economy, worry about health (health anxiety), maladaptive mental and behavioral coping, and negative and positive metacognitions as constant covariates will be added, together with the interactions of these constant covariates with time. These interactions represent tests of H2 about the covariates predicting change in loneliness. Finally, the T2 levels of worry about job and/or economy, worry about health (health anxiety), maladaptive mental and behavioral coping, and negative and positive metacognitions as constant covariates will be added, together with the interactions of these constant covariates with time. These interactions represent tests of H2 about the change in the covariates from T1 to T2 predicting change in loneliness from T1 to T2.

To analyze the influence of level and change in loneliness on change in depression and anxiety (H3), depression and anxiety are used as dependent variables in two mixed models, with first the interaction of time with loneliness at T1 and then the interaction of time with loneliness at T2 as covariates. The main effects of these variables are included as well as all significant terms from the analyses of loneliness as dependent variable.

Reliable change in loneliness will be assessed using the formula of Jacobson and Truax (1991). The statistical analyses were done in the program SPSS 25.0 (IBM Corp, 2018).

Sensitivity analyses Sensitivity analyses will be conducted after selecting a random sample of participants to reflect the proportion of subgroups in the Norwegian adult population.

ELIGIBILITY:
Inclusion Criteria:

* all adults residing in Norway

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Eligible participants are all individuals of 18 years and above, who are living in Norway and thus experience identical distancing protocols, and who provide informed consent to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 10084 (Estimated)
Dates: Start 2020-06-22 (Estimated); Primary Completion 2020-07-13 (Estimated); Study Completion 2020-07-13 (Estimated)

PRIMARY OUTCOMES:
UCLA Loneliness Scale-8 (ULS-8) | From 22nd of June to 13th of July
  The UCLA Loneliness Scale-8 (ULS-8; Hays & DiMatteo, 1987) measures the frequency and intensity of aspects of the lonely experience, using a 1 (never), 2 (rarely), 3 (sometimes) and 4 (often) scale. A composite score is computed by summing the items after reverse coding when appropriate, with composites ranging from 8 to 32. A score greater than half the maximum score (16) has been used to indicate caseness (Shevlin, Murphy, Mallett, Stringer, & Murphy, 2013). This implies that respondents at least sometimes experience at least one of the loneliness aspects described in the 8 items. The ULS-8 has demonstrated good psychometric properties (Hays & DiMatteo, 1987; Hartshorne, 1993).
Patient Health Questionnaire-9 (PHQ-9) | From 22nd of June to 13th of July
  The Patient Health Questionnaire-9 (PHQ-9; Kroenke, Spitzer, & Williams, 2001) consists of nine items covering the DSM-IV criteria for major depression scored on a four-point 0 (not at all) to 3 (almost every day) scale, with total scores ranging from 0 to 27. The PHQ-9 has revealed good psychometric properties, as demonstrated by Kroenke, Spitzer, and Williams (2001).
Generalized Anxiety Disorder-7 (GAD-7) | From 22nd of June to 13th of July
  The Generalized Anxiety Disorder-7 (GAD-7; Kroenke, Spitzer, Williams, Monahan & Löwe, 2007) consists of seven items covering the DSM-IV criteria for GAD scored on a four-point 0 (not at all) to 3 (almost every day) scale, with total scores ranging from 0 to 21. The GAD-7 has revealed construct validity and reliability (Kroenke et al., 2007; Löwe et al., 2008).

CONTACTS AND LOCATIONS:
Overall Officials: Omid Ebrahimi, Cand Psychol, Principal Investigator — University of Oslo and Modum Bad; Asle Hoffart, PhD, Principal Investigator — Modum Bad and University of Oslo; Sverre Urnes Johnson, PhD, Principal Investigator — University of Oslo and Modum Bad

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hoffart A, Johnson SU, Ebrahimi OV. Loneliness during the COVID-19 pandemic: change and predictors of change from strict to discontinued social distancing protocols. Anxiety Stress Coping. 2022 Jan;35(1):44-57. doi: 10.1080/10615806.2021.1958790. Epub 2021 Jul 27. PMID 34314285